CLINICAL TRIAL: NCT01427127
Title: Effect of Ramosetron on Bowel Motility and PONV After Laparoscopic Stomach and Colorectal Resection
Brief Title: Effect of Ramosetron on Bowel Motility After Colorectal Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Mi Kyeong Kim, Assistant Professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RAMS
Record Dates: First submitted 2011-08-25; First posted 2011-09-01 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — ramosetron

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ramosetron (Experimental): Patients received intravenous ramosetron 0.3 mg at the end of surgery and 24hr after surgery.
  Interventions: Drug: Ramosetron
- Normal saline (Placebo Comparator): Patients received intravenous normal saline at end of surgery and 24hr after surgery.
  Interventions: Drug: Ramosetron

INTERVENTIONS:
Drug: Ramosetron — Patients received intravenous ramosetron 0.3 mg at end of surgery and 24hr after surgery.
  Other Names: nasea (Astellas Pharma Korea, Inc.)

SUMMARY:
Ramosetron is effective in preventing postoperative nausea and vomiting. Several studies reported that ramosetron is also effective treatment diarrhea-predominant irritable bowel syndrome. The investigators examine the effect of ramosetron used for preventing postoperative nausea and vomiting on bowel motility.

DETAILED DESCRIPTION:
Ramosetron, a new potent and long-acting selective 5-HT3 receptor antagonist, is effective for preventing postoperative nausea and vomiting. Also several studies reported that ramosetron is effective treatment of irritable bowel syndrome because it inhibits the accelerated colonic transit, abnormal colonic water transport, defecation abnormality, and the lowered colonic perceptual threshold by corticotrophin-releasing hormone. There is no study about the effect of ramosetron used for preventing postoperative nausea and vomiting on postoperative bowel motility. In this study, the investigators examine the effect of ramosetron on postoperative bowel motility.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 yr of age,
* ASA I or II,
* scheduled for laparoscopic colorectal surgery

Exclusion Criteria:

* antiemetic use within 24hr prior to surgery
* steroid use within 24hr prior to surgery or 48hr after surgery
* insulin dependent DM
* cardiovascular or pulmonary disease
* renal or hepatic insufficiency
* BMI >=35kg/m2
* pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
time from surgery to passage of gas | within 10days after surgery
time from surgery to defecation | within 10 days after surgery

SECONDARY OUTCOMES:
incidence and severity of postoperative nausea and vomiting | 0 - 6 hours, 6-24 hours, and 24-48 hours after surgery
  incidence: number of patients who experienced postoperative nausea and vomiting severity: verbal rating scale (VRS, 11 point scale) 0= no nausea to 10 = worst possible nausea

CONTACTS AND LOCATIONS:
Overall Officials: Mi Kyeong Kim, Principal Investigator — School of Medicine, Kyung Hee University
Locations (1):
- School of Medicine, Kyung Hee University, Seoul, South Korea